CLINICAL TRIAL: NCT06061770
Title: Comparison of the Effectiveness of an Adapted Physical Activity Program in a Dedicated Structure to a Self-program in Patients in Chronic Phase of a Stroke
Acronym: StrokAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCAPHM21_0439
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First APA program (Experimental): The evaluation of the primary endpoint to meet our main objective will be done at W13 for both groups. The addition of an APA program in autonomy following the structured program for group 1 will make it possible to answer a secondary question focusing on the comparison of the effectiveness of the self-directed program carried out alone or following a structured program.
  1st group: D0: Include S1-S12: APA program at IUR Valmante S13: Break S14-S25: APA Autoprogram
  In addition, the patients in group 1 are maintained in the follow-up to study the maintenance of any observed effect.
  Interventions: Other: Adapted physical activity program
- Second APA program (Active Comparator): Our study design provides for compensatory participation in the structured program for patients in group 2, following the self-program. From an ethical point of view, this scheme allows all patients included in the structured APA program to benefit.
  2nd group: D0: Include S1-S12: APA Autoprogram S13: End of study S14-S25: APA program at IUR Valmante compensatory
  Interventions: Other: Adapted physical activity self-program

INTERVENTIONS:
Other: Adapted physical activity program — Rehabilitation
  Arms: First APA program
Other: Adapted physical activity self-program — Rehabilitation
  Arms: Second APA program

SUMMARY:
This is a prospective, randomized, controlled, two parallel arms, single-blind pilot study. In this design, all included patients in the chronic phase of a stroke will receive both modes of physical activity.

This study includes patients over 18 years of age with spastic hemiparesis sequelae of a first unilateral hemispheric stroke older than 6 months and able to walk for 6 minutes. The non-inclusion criteria were the inability to walk without human assistance (with or without technical aids), the existence of cognitive disorders compromising informed consent, in particular the inability to understand the objective and the modalities of the protocol, the inability to communicate with the examiners, and the presence of an additional neurological disorder or a pathology contraindicating the practice of physical activity.

The primary endpoint is based on daily activity measurement by measuring the number of steps per day, collected over the duration of the study, via a Stepwatch™ device. Secondary end points involve a written physical activity report, assessment of walking ability (via walking-test 6, heart rate, and blood pressure), a measure of perceived exertion, stroke-specific quality of life, balance, and motivation to perform physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Left or right spastic hemiparesis after a first hemorrhagic or ischemic unilateral stroke older than 6 months
* Walking possible for 6 minutes

Exclusion Criteria:

* Inability to walk without human assistance (with or without technical aids)
* Cognitive impairment that compromises informed consent, including inability to understand the purpose and terms of the protocol
* Inability to communicate
* Presence of an additional neurological disorder
* Medical conditions that contraindicate physical activity, such as an unbalanced cardiovascular or respiratory condition
* Concurrent participation in another clinical research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
Daily activity measurement | through study completion
  Measuring the number of steps per day, collected over the duration of the study, via a Stepwatch device

SECONDARY OUTCOMES:
the rate physical activities in Written report | through study completion
  carried out by the patient, more or less helped by his close entourage, recorded in a notebook given at the beginning of the study
6-minute walk test (6MWT) | at inclusion Day and at the 13th week (and the 26th week for one group only)
  A test validated in the literature that consists of measuring the greatest distance that a subject can travel on a flat surface (30 meter corridor) in 6 minutes.
Measurement of heart rate at rest and after 6-minute walk test | at inclusion Day and at the 13th week (and the 26th week for one group only)
  with a blood pressure cuff
Measurement of systolic blood pressure at rest and after 6-minute walk test | at inclusion Day and at the 13th week (and the 26th week for one group only)
  with a blood pressure cuff
Borg Rating Scale of Exertion | at inclusion Day and at the 13th week (and the 26th week for one group only)
  test validated in the literature that allows the evaluation of the perception of effort by the patient ; minimum value : 0 = rest : no exertion ; maximum value : 10 = maximal exertion
Stroke Specific Quality of Life scale (SS-QoL) | at inclusion Day and at the 13th week (and the 26th week for one group only)
  A test validated in French in the literature that assesses the specific quality of life of stroke patients in 49 items ; minimum value : 1 = Total help/ Couldn't do it at all/ Strongly agree ; maximum value : 5 = No help needed/ No trouble at all/ Strongly disagree
Berg Balance Scale (BBS) | at inclusion Day and at the 13th week (and the 26th week for one group only)
  validated scale allowing, by means of 14 instructions, an evaluation of balance, reproducible and sensitive to change ; minimum score : 0-20 = high risk of falling ; maximal score : 56 = no risk of falling
Activity-specific Balanced Confidence scale (ABC scale) | at inclusion Day and at the 13th week (and the 26th week for one group only)
  French language validated scale assessing the patient's confidence in his or her balance, using 16 situations where the subject is asked to rate his or her balance on a numerical scale ; minimal rate : 0% = not at all confident ; maximal rate : 100% = completely confident
Behavioral regulation in exercise questionnaire | at inclusion Day and at the 13th week (and the 26th week for one group only)
  scale used in the literature to assess motivation to perform physical activity ; minimal value : 1 = not true at all ; maximal value : 7 = absolutely true

CONTACTS AND LOCATIONS:
Locations (1):
- Médecine Physique et de Réadaptation, CHU Hôpital Sainte Marguerite, Marseille, Bouches du Rhône, France

IPD SHARING:
Plan to Share IPD: Yes
Data sharing statements that meet these ICMJE requirements Individual pseudonymous data of participants may be available The data that may be shared are the individual data of the participants which underlie the results reported in this article, after de-identification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: For researchers who provide a methodologically sound proposal. Types of analyses: Achieve the objectives of the approved proposal. Proposals should be sent to maeva.cotinat@ap-hm.fr

REFERENCES:
- [Derived] Satger E, Prieur-Blanc N, Viton JM, Auquier P, Bensoussan L, Cotinat M. Effectiveness of an institution-based adapted physical activity programme versus a home-based self-management programme for chronic poststroke adults: protocol for a randomised controlled study. BMJ Open. 2024 Jul 20;14(7):e084688. doi: 10.1136/bmjopen-2024-084688. PMID 39032927